CLINICAL TRIAL: NCT00423293
Title: A Phase II Evaluation of Dose-Painted Intensity-Modulated Radiation Therapy (IMRT) in Combination With 5-Fluorouracil (5-FU) and Mitomycin-C for Reduction of Acute Morbidity in Carcinoma of the Anal Canal
Brief Title: Intensity-Modulated Radiation Therapy, Fluorouracil, and Mitomycin C in Treating Patients With Invasive Anal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0529; CDR0000524057
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Anal Cancer
Keywords: stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; basaloid carcinoma of the anus; cloacogenic carcinoma of the anus; squamous cell carcinoma of the anus
MeSH Terms: conditions — Anus Neoplasms; Anal Canal Carcinoma | interventions — Fluorouracil; Mitomycin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-FU + Mitomycin + IMRT (Other): 5-FU + Mitomycin + IMRT
  Interventions: Drug: fluorouracil; Drug: mitomycin C; Radiation: Intensity-modulated radiation therapy

INTERVENTIONS:
Drug: fluorouracil — 1000 mg/m^2/day 96-hour continous infusion (M-F) starting on day 1 and again on day 29 of radiation therapy.
Drug: mitomycin C — 10 mg/m^2 intravenous therapy on day 1 and day 29 of radiation therapy.
Radiation: Intensity-modulated radiation therapy — Prescription dose depends on tumor staging.
  T2N0: The primary tumor PTV (planning target volume) (PTVA) receives 50.4 Gy in 28 fractions (fx) at 1.8 Gy/fx. The nodal PTVs receive 42 Gy in 28 fx at 1.5 Gy/fx. PTVA receive 50.4 Gy in 28 fractions at 1.8 Gy/fx. PTV42 receive 42 Gy in 28 fx at 1.5 Gy/fx and will include all nodal regions.
  T3N0 or T4N0: The primary tumor PTV (PTVA) will receive 54 Gy in 30 fx at 1.8 Gy/fx. The nodal PTVs will receive 45 Gy in 30 fx at 1.5 Gy/fx. PTVA will receive 54 Gy in 30 fx at 1.80 Gy/fx. PTV45 will receive 45 Gy in 30 fx electively at 1.5 Gy/fx and will include all nodal regions.
  For N+ disease: The primary tumor PTV (PTVA) will receive 54 Gy in 30 fx at 1.8 Gy/fx. For involved nodes ≤ 3 cm in maximum dimension, the involved nodal PTV will receive 50.4 Gy in 30 fx at 1.68 Gy/fx. For involved nodes > 3 cm in maximum dimension, the involved nodal PTV will receive 54 Gy in 30 fx at 1.80 Gy/fx.

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as fluorouracil and mitomycin C, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with 5-fluorouracil (5-FU) and mitomycin C may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving intensity-modulated radiation therapy together with fluorouracil and mitomycin C works in treating patients with invasive anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if dose-painted, intensity-modulated radiation therapy (IMRT), fluorouracil, and mitomycin C decreases the combined rate of gastrointestinal and genitourinary adverse events (grade II or greater) by at least 15% in the first 90 days after the start of treatment in patients with primary invasive carcinoma of the anal canal compared to patients treated on the radiotherapy, fluorouracil, and mitomycin C arm on clinical trial RTOG 98-11.

Secondary

* Determine the feasibility of performing IMRT in these patients in a cooperative group setting.
* Evaluate adverse events experienced by patients treated with this regimen and to decrease the grade 2 and higher and grade 3 and higher overall adverse event rates by 15% or 20% as compared to the radiotherapy and mitomycin C arm of RTOG 98-11.
* Evaluate the total duration of radiotherapy.
* Evaluate the efficacy of this regimen, in terms of locoregional failure, disease-free survival, time to colostomy, colostomy-free survival, and overall survival of these patients.
* Determine clinical complete response at 8 weeks after completion of study treatment.

OUTLINE: This is a multicenter study.

Patients receive mitomycin C IV over 10-30 minutes on days 1 and 29 and fluorouracil IV continuously over 96 hours on days 1-4 and 29-32. Patients also undergo dose-painted intensity-modulated radiation therapy once daily, 5 days a week, for 5½ to 6 weeks beginning on day 1. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 59 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the anal canal, including any of the following subtypes:

  * Squamous cell
  * Basaloid
  * Cloacogenic
* Primary invasive disease
* T2-4, N0-3 disease

  * Clinically positive small inguinal nodes (i.e., < 1 cm in size) must be confirmed by biopsy (preferably fine-needle aspiration) within the past 6 weeks
  * Biopsy is not required for enlarged inguinal, perirectal, or pelvic nodes on exam or CT scan that are found to be ≥ 1.0 cm and are considered to be clinically positive

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Hemoglobin ≥ 8.0 g/dL (transfusion or other intervention allowed)
* ALT and AST < 3 times upper limit of normal
* Absolute neutrophil count ≥ 1,800/mm³
* Serum creatinine ≤ 1.5 mg/dL
* Platelet count ≥ 100,000/mm³
* Bilirubin < 1.4 mg/dL
* WBC ≥ 3,000/mm³
* INR ≤ 1.5
* No known AIDS

  * HIV-positive patients without AIDS are eligible
  * HIV test required for patients with clinical suspicion of AIDS
* No other invasive malignancy within the past 3 years except for nonmelanomatous skin cancer
* No severe, active comorbidity, defined as any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring IV antibiotics
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study treatment
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Uncontrolled diabetes mellitus, uncompensated heart disease, and/or uncontrolled high blood pressure, that in the opinion of the patient's treating physician, requires an immediate change in management

    * Patients may be eligible if appropriate changes in management have resulted in adequate control of the above mentioned conditions
  * Other immunocompromised status (e.g., organ transplantation or chronic glucocorticoid use)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiation therapy to the pelvis that would result in overlap of radiation therapy fields
* No prior systemic chemotherapy for cancer of the anus
* No prior surgery for cancer of the anus that removed all macroscopic anal cancer
* No concurrent sargramostim (GM-CSF)
* No concurrent amifostine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Kachnic, MD, Study Chair — Boston Medical Center
Locations (172):
- United States (169):
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Solano Radiation Oncology Center, Vacaville, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital, Boca Raton, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Bay Medical, Panama City, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - St. Vincent Oncology Center, Indianapolis, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - Saint Louis, St Louis, Missouri
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center Dallas Southwest, Dallas, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Harrison Medical Center, Bremerton, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
- Canada (3):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5-FU + Mitomycin + IMRT
Started | 63
Completed | 52 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 11
Not completed — Ineligible / No protocol treatment | 11

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 58 [34 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Acute Gastrointestinal (GI) and Genitourinary (GU) Adverse Events (AE) ≥ Grade 2 as Defined by CTCAE v3.0 (Common Terminology Criteria for Adverse Events)
Description: Highest grade adverse event per subject were counted. Adverse events were graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Acute toxicities occur within 90 days of the start of treatment.
Time Frame: From the start of treatment to 90 days
Population: Eligible patients with adverse event information.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants | 77 [NA to 87] — This is a one-sided confidence interval.
Statistical Analysis 1: Comparison: 5-FU + Mitomycin + IMRT; The RT+ 5-FU + Mitomycin-C arm on previous Radiation Therapy Oncology Group (RTOG) study 9811 [NCT00003596] had a 77% rate of >= grade 2 GI and GU adverse events. The null hypothesis for this study design was a 15% reduction for that rate. Fifty-four evaluable patients provides 80% power to detect a 15% reduction, using a one-sided chi-squared test with a type I error rate of 0.05. (With 52 patients, the power is reduced to 78%.); Test type: Superiority or Other; p = 0.50, Chi-squared — One-sided p-value comparing to a rate of 78% (the historical rate was updated after the study design)

2. Secondary Outcome: Number of Patients With Major Radiation Planning Deviations
Description: Deviations in intensity-modulated radiation therapy technique (IMRT) planning were determined by central review by the radiation oncology co-chairs of the study.
Time Frame: Planning occurred prior to radiation therapy
Population: All eligible patients who started IMRT
Measure: Count of Participants; unit: Participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 51
Participants | 0

3. Secondary Outcome: Percentage of Subjects With Acute Adverse Events (AE)
Description: as for outcome 1
Time Frame: From the start of treatment to 90 days
Population: Eligible patients who started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants
  GI Grade 2+ | 73 [NA to 83] — One-sided confidence interval
  GU Grade 2+ | 15 [NA to 28] — One-sided confidence interval
  Hematologic Grade 2+ | 73 [NA to 83] — One-sided confidence interval
  Skin Grade 2+ | 75 [NA to 85] — One-sided confidence interval
  Any Grade 2+ | 94 [NA to 99] — One-sided confidence interval
  Any Grade 3+ | 83 [NA to 91] — One-sided confidence interval
Statistical Analysis 1: Comparison: 5-FU + Mitomycin + IMRT; Percentage of patients with GI grade 2+ adverse events were compared to the historical rate of 73%. Null hypothesis: same or greater than historical rate. Alternative hypothesis: less than historical rate; Test type: Superiority; p = 0.5, Chi-squared; One-sided significance level = 0.05
Statistical Analysis 2: Comparison: 5-FU + Mitomycin + IMRT; Percentage of patients with GU grade 2+ adverse events were compared to the historical rate of 20%. Null hypothesis: same or greater than historical rate. Alternative hypothesis: less than historical rate; Test type: Superiority; p = 0.18, Chi-squared; One-sided significance level = 0.05
Statistical Analysis 3: Comparison: 5-FU + Mitomycin + IMRT; Percentage of patients with hematologic grade 2+ adverse events were compared to the historical rate of 85%. Null hypothesis: same or greater than historical rate. Alternative hypothesis: less than historical rate; Test type: Superiority; p = 0.032, Chi-squared; One-sided significance level = 0.05
Statistical Analysis 4: Comparison: 5-FU + Mitomycin + IMRT; Percentage of patients with skin grade 2+ adverse events were compared to the historical rate of 83%. Null hypothesis: same or greater than historical rate. Alternative hypothesis: less than historical rate; Test type: Superiority; p = 0.10, Chi-squared; One-sided significance level = 0.05
Statistical Analysis 5: Comparison: 5-FU + Mitomycin + IMRT; Percentage of patients with any grade 2+ adverse events were compared to the historical rate of 98%. Null hypothesis: same or greater than historical rate. Alternative hypothesis: less than historical rate; Test type: Superiority; p = 0.12, Chi-squared; One-sided significance level = 0.05
Statistical Analysis 6: Comparison: 5-FU + Mitomycin + IMRT; Percentage of patients with any grade 3+ adverse events were compared to the historical rate of 87%. Null hypothesis: same or greater than historical rate. Alternative hypothesis: less than historical rate; Test type: Superiority; p = 0.23, Chi-squared; One-sided significance level = 0.05

4. Secondary Outcome: Percentage of Subjects With Late Adverse Events (AE)
Description: Highest grade adverse event per subject were counted. Adverse events were graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Late toxicities occur greater than 90 days from the start of treatment.
Time Frame: From 91 days after start of study treatment to the end of follow-up. Maximum follow-up at time of analysis was 9.2 years.
Population: Eligible patients who started IMRT and were on-study > 90 days from the start of treatment (or did not withdraw consent until after 90 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 51
percentage of participants
  GI/GU Grade 2+ | 35 [24 to 49]
  Non-Hematologic Grade 2+ | 67 [53 to 78]
  Any Grade 2+ | 75 [61 to 81]
  Any Grade 3+ | 20 [11 to 33]

5. Secondary Outcome: Clinical Complete Response Rate
Description: A complete clinical response was defined as complete resolution of all palpable tumor determined by digital rectal exam and proctosigmoidoscopy supplemented with pelvic axial imaging.
Time Frame: 8 and 12 weeks after treatment completion (corresponding to 14 and 18 weeks from registration)
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants
  8 weeks after treatment | 64 [50 to 75]
  12 weeks after treatment | 81 [68 to 89]

6. Secondary Outcome: Duration of Radiotherapy Treatment
Description: Number of days from radiotherapy treatment start to radiotherapy treatment end
Time Frame: From start to end of radiation therapy (6 weeks)
Population: Eligible patients who started IMRT
Measure: Median (Full Range); unit: Days
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 51
Days | 43 [32 to 59]

7. Secondary Outcome: Five-year Rate of Overall Survival
Description: Overall survival time is defined as time from registration/randomization to the date of death from any cause. Overall survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From registration to 5 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants | 76 [61 to 86]

8. Secondary Outcome: Five-year Rate of Disease-free Survival
Description: Disease-free survival time is defined as time from registration to the date of local-regional failure, the appearance of distant metastases, the appearance of a second primary failure, or date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive without failure are censored at the date of last contact. Local failure is defined as any measurable disease after 12 weeks from the completion of chemoradiation therapy. Local failure is defined as: a) For patients with no disease in pelvic and/or groin nodes, the appearance of disease in pelvic or groin nodes; b) For patients with disease in pelvic and/or groin nodes at study entry, nodal recurrence following clearance or persistent nodal disease for more than 12 weeks after completion of treatment.
Time Frame: From registration to 5 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants | 70 [56 to 81]

9. Secondary Outcome: Five-Year Cumulative Incidence Rate of Local-regional Failure
Description: Local-regional failure time is defined as time from registration to date of failure and is estimated by the cumulative incidence method. Patients last known to be alive without failure are censored at the date of last contact. Local-regional failure is defined as a local or regional failure. Local failure is defined as any measurable disease after 12 weeks from the completion of chemoradiation therapy. Regional failure is defined as: a) For patients with no disease in pelvic and/or groin nodes, the appearance of disease in pelvic or groin nodes; b) For patients with disease in pelvic and/or groin nodes at study entry, nodal recurrence following clearance or persistent nodal disease for more than 12 weeks after completion of treatment.
Time Frame: From registration to 5 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants | 16 [7 to 27]

10. Secondary Outcome: Five-Year Cumulative Incidence Rate of Distant Failure
Description: Distant failure time is defined as time from registration to the appearance of distant metastases and is estimated by the cumulative incidence method. Patients last known to be alive without failure are censored at the date of last contact.
Time Frame: From registration to 5 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants | 16 [7 to 27]

11. Secondary Outcome: Five-Year Cumulative Incidence Rate of Colostomy Failure
Description: Colostomy failure time is defined as time from registration to the date of colostomy or abdominoperineal (A-P) resection and is estimated by the cumulative incidence method. Patients last known to be alive without failure are censored at the date of last contact.
Time Frame: From registration to 5 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants | 10 [4 to 20]

12. Secondary Outcome: Five-Year Rate of Colostomy-free Survival
Description: Colostomy-free survival time is defined as time from registration to date of colostomy or abdominoperineal (A-P) resection, or date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive without failure are censored at the date of last contact.
Time Frame: From registration to 5 years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-FU + Mitomycin + IMRT
Number analyzed (Participants) | 52
percentage of participants | 74 [59 to 84]

ADVERSE EVENTS:
Description: Eligible patients with adverse event data are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | 5-FU + Mitomycin + IMRT
Serious Adverse Events (participants affected / at risk) | 6/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU + Mitomycin + IMRT (N=52)
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Cystitis noninfective (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-FU + Mitomycin + IMRT (N=52)
Anemia (Blood and lymphatic system disorders) | 35
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 13
Anal fistula (Gastrointestinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 5
Anal pain (Gastrointestinal disorders) | 15
Anal stenosis (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Colonic hemorrhage (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 18
Diarrhea (Gastrointestinal disorders) | 42
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 3
Esophageal pain (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 6
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 25
Nausea (Gastrointestinal disorders) | 28
Oral pain (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 16
Rectal hemorrhage (Gastrointestinal disorders) | 14
Rectal pain (Gastrointestinal disorders) | 10
Rectal ulcer (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Chills (General disorders) | 1
Death NOS (General disorders) | 1
Edema limbs (General disorders) | 7
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 33
Fever (General disorders) | 4
General disorders and administration site conditions - Other (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pain (General disorders) | 7
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 2
Allergic reaction (Immune system disorders) | 2
Bladder infection (Infections and infestations) | 3
Infections and infestations - Other (Infections and infestations) | 7
Lung infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 31
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 9
Vascular access complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 2
CD4 lymphocytes decreased (Investigations) | 1
CPK increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 2
Investigations - Other (Investigations) | 6
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 33
Platelet count decreased (Investigations) | 32
Weight loss (Investigations) | 12
White blood cell decreased (Investigations) | 33
Anorexia (Metabolism and nutrition disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 12
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 19
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 13
Hyponatremia (Metabolism and nutrition disorders) | 16
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 4
Nervous system disorders - Other (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 8
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 6
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 4
Libido decreased (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 8
Hematuria (Renal and urinary disorders) | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 5
Urinary frequency (Renal and urinary disorders) | 18
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 4
Urine discoloration (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 2
Penile pain (Reproductive system and breast disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 9
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 4
Scrotal pain (Reproductive system and breast disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 6
Vaginal hemorrhage (Reproductive system and breast disorders) | 2
Vaginal inflammation (Reproductive system and breast disorders) | 2
Vaginal obstruction (Reproductive system and breast disorders) | 5
Vaginal pain (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 12
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2
Skin atrophy (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 12
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Skin induration (Skin and subcutaneous tissue disorders) | 4
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No